CLINICAL TRIAL: NCT04201600
Title: Relations of Glucose Variability with Cognitive Function and Functional Status Among Older Adults At Risk for Diabetes
Brief Title: Glucose Variability and Cognition in Prediabetes
Status: Recruiting | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Baltimore VA Medical Center (U.S. Federal Agency); University of Maryland, Baltimore County (Other)
Responsible Party: Principal Investigator, Leslie Katzel, Associate Professor, University of Maryland, Baltimore
Other Study IDs: HP-00087044
Record Dates: First submitted 2019-12-05; First posted 2019-12-17 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Glucose Metabolism Disorders (Including Diabetes Mellitus); Cognitive Decline; Functional Status; PreDiabetes; Aging; Depression
Keywords: Glucose Variability; Continuous Glucose Monitoring System (CGMS); Prediabetes; Aging; Physical Functioning; Neurocognition; Cognitive Decline
MeSH Terms: conditions — Glucose Metabolism Disorders; Cognitive Dysfunction; Prediabetic State; Depression | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples, inflammatory markers, fasting glucose
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Middle-aged and Older adults with Prediabetes: Middle-aged and Older adults with Prediabetes
  Interventions: Device: Continuous Glucose Monitoring System (CGMS)

INTERVENTIONS:
Device: Continuous Glucose Monitoring System (CGMS) — Continuous Glucose Monitoring System (CGMS)- minimally invasive sensors that measure glucose concentrations at 5-min intervals over several days.

SUMMARY:
This study examines the association of variability in glucose values over a 10-day period with cognitive function and functional status among individuals with prediabetes, aged 50 or older.

DETAILED DESCRIPTION:
Type 2 diabetes (T2DM) is now widely considered a major public health epidemic. T2DM is highly prevalent worldwide, is among the leading causes of death, and is an independent risk factor for dementia and less severe forms of cognitive dysfunction. The investigators are utilizing novel technology to understand the role of variability in glucose on neurocognition and functional status among middle-aged and older adults at risk for diabetes. The central hypothesis is that even before diabetes onset, variability in glucose will be associated with worse cognitive function and lower functional status. Participants will be asked to wear a glucose monitoring device over a 10-day period in their home environment. Assessment of functional status and neurocognitive function, in addition to sociodemographic factors, health habits and mood will also occur over two study visits.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 years and older
* At least 8th grade education

Exclusion Criteria:

* Diagnosed type 1 or type 2 diabetes
* Current use of mediation for diabetes (oral hypoglycemic agents, insulin), or with diabetic properties (e.g., steroids)
* Chronic disorders (cardiovascular disease, peripheral vascular disease, stroke, transient ischemic attack, chronic kidney disease, past year cancer)
* Neurological disorders (e.g., Parkinson's, epilepsy, multiple sclerosis)
* History of dementia or suspected dementia
* Known HIV
* Serious mental illness, psychosis, or use of psychotropic medication
* Heavy alcohol use

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults aged 50 years and older with prediabetes of any duration
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Aggregate Executive Functioning Score | Day 10
  Scores on the following standard neurocognitive tests will be z-transformed based on their respective means and standard deviations and combined into one aggregate total score such that higher values mean better executive functioning:
  Trails Making A and B, The Stroop-Color Word Test, Digit Span subscale of the Wechsler Adult Intelligence Scale - Revised (WAIS-IV), Digit Symbol Substitution Test (DSST)
Aggregate Memory Score | Day 10
  Scores on the following standard neurocognitive tests will be z-transformed based on their respective means and standard deviations and combined into one aggregate total score such that higher values mean better memory ability:
  California Verbal Learning Test, Benton Visual Retention Test
Aggregate Language Score | Day 10
  Scores on the following standard neurocognitive tests will be z-transformed based on their respective means and standard deviations and combined into one aggregate total score such that higher values mean better language abilities:
  Boston Naming Test, Controlled Oral Word Association Test (COWA)

SECONDARY OUTCOMES:
Aggregate Physical Functioning Score | Day 10
  Scores on the following standard neurocognitive tests will be summed into one aggregate total score such that higher values mean better physical functioning:
  gait speed, short physical performance battery (SPPB), handgrip strength, and four-square step test
Activities of Daily Living (ADL) total score | Day 10
  Responses on this standard measure will be scored according to guidelines to create a total score for functional status
Instrumental Activities of Daily Living (IADL) total score | Day 10
  Responses on this standard measure will be scored according to guidelines to create a total score for functional status

CONTACTS AND LOCATIONS:
Overall Officials: Tasneem Khambaty, PhD, Principal Investigator — University of Maryland, Baltimore County
Locations (1):
- Baltimore VA Geriatric Research Education and Clinical Center (GRECC), Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No